CLINICAL TRIAL: NCT02841488
Title: Comparative Study Between Systemic Analgesia and Continuous Sciatic Nerve Block in Patients With Chronic Obstructive Arterial Disease and Ischemic Pain in Lower Limbs
Brief Title: Ischemic Pain Control With Analgesic Methods Clinical Trial
Acronym: ISCHAEMIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, M.D., University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 55187516.4.0000.0068
Record Dates: First submitted 2016-07-17; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Arterial Occlusive Diseases
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — Fentanyl; Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous nerve block (Active Comparator): Continuous peripheral sciatic nerve block through popliteal perineural catheter with ropivacaine
  Interventions: Procedure: Continuous peripheral sciatic nerve block; Drug: Ropivacaine; Device: Perineural catheter
- Systemic analgesia (Active Comparator): Intravenous fentanyl patient controlled analgesia device
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Procedure: Continuous peripheral sciatic nerve block — Continuous infusion of local anesthetics through perineural sciatic nerve catheter
  Other Names: Perineural sciatic catheter
  Arms: Continuous nerve block
Drug: Fentanyl — Use of patient controlled analgesia device with intravenous fentanyl
  Other Names: Intravenous fentanyl
  Arms: Systemic analgesia
Drug: Ropivacaine
  Arms: Continuous nerve block
Device: Perineural catheter
  Arms: Continuous nerve block

SUMMARY:
This project is one of four components of a thematic project that aims to evaluate the use of ultrasound in regional blocks, called "Use of ultrasound in regional blocks and injections for the treatment of acute and chronic pain."

It will evaluate quantitative and qualitative control of ischemic pain in the lower limbs in patients with peripheral arterial occlusive disease through continuous sciatic nerve block by perineural catheter, popliteal approach, compared to systemic analgesia based on opioids.

DETAILED DESCRIPTION:
BACKGROUND: Peripheral arterial occlusive disease (PAOD) commonly evolves with intense ischemic pain in the lower limbs, which is hard to control with systemic analgesics, and continuous regional anesthesia may be an alternative, with adequate analgesia and lower incidence of side effects.

OBJECTIVES: evaluate qualitative and quantitative pain control, incidence of adverse effects and operative results in patients with PAOD undergoing continuous anesthetic blockade of the sciatic nerve by perineural catheter compared to systemic analgesia based on opioids and adjuvant medications.

METHODS: It is a randomized clinical trial, covered for evaluators. It will include 56 patients with PAOD Fontaine IV, with pain by the presence of ulcerations located on foot. A group will be submitted to continuous regional anesthesia of sciatic nerve through perineural catheter and another group will have its pain control through patient controlled analgesia device with intravenous fentanyl. The primary dependent variable will be pain, through the numerical pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old who have strong or moderate persistent ischemic pain in the lower limbs, due to peripheral artery occlusive disease, classified as Fontaine IV (pain at rest and presence of ulcer or gangrene).

Exclusion Criteria:

* Uncooperative patients, coagulation disorders, patients with liver failure, who have atrioventricular block second or third degree, who refuse to be submitted to peripheral nerve block, with systemic or procedure site local infection infection, peripheral or central neuropathy history, allergies to local anesthetics or to any of the drugs to be used in the study and difficulty in understanding the use of the PCA (patient-controlled analgesia) device and evaluation methods used in the study .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | up to 28th day
  Verbal numerical scale

SECONDARY OUTCOMES:
Opioids Adverse effects | up to 28th day
  Nausea, vomiting, constipation, sedation

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim E Vieira, PhD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Selvin E, Erlinger TP. Prevalence of and risk factors for peripheral arterial disease in the United States: results from the National Health and Nutrition Examination Survey, 1999-2000. Circulation. 2004 Aug 10;110(6):738-43. doi: 10.1161/01.CIR.0000137913.26087.F0. Epub 2004 Jul 19. PMID 15262830
- [Background] Navas-Acien A, Selvin E, Sharrett AR, Calderon-Aranda E, Silbergeld E, Guallar E. Lead, cadmium, smoking, and increased risk of peripheral arterial disease. Circulation. 2004 Jun 29;109(25):3196-201. doi: 10.1161/01.CIR.0000130848.18636.B2. Epub 2004 Jun 7. PMID 15184277
- [Background] Belch JJ, Topol EJ, Agnelli G, Bertrand M, Califf RM, Clement DL, Creager MA, Easton JD, Gavin JR 3rd, Greenland P, Hankey G, Hanrath P, Hirsch AT, Meyer J, Smith SC, Sullivan F, Weber MA; Prevention of Atherothrombotic Disease Network. Critical issues in peripheral arterial disease detection and management: a call to action. Arch Intern Med. 2003 Apr 28;163(8):884-92. doi: 10.1001/archinte.163.8.884. No abstract available. PMID 12719196
- [Background] McDaniel MD, Cronenwett JL. Basic data related to the natural history of intermittent claudication. Ann Vasc Surg. 1989 Jul;3(3):273-7. doi: 10.1016/S0890-5096(07)60040-5. No abstract available. PMID 2673321
- [Background] Marquis P, Lecasble M, Passa P. [Quality of life of patient with peripheral arterial obliterative disease treated with ifenprodil tartrate. Results of an ARTEMIS study]. Drugs. 1998;56 Suppl 3:37-48. doi: 10.2165/00003495-199856003-00005. French. PMID 9844701
- [Background] Campbell WB, Marriott S, Eve R, Mapson E, Sexton S, Thompson JF. Anaesthesia and analgesia for major lower limb amputation. Cardiovasc Surg. 2000 Dec;8(7):572-5. doi: 10.1016/s0967-2109(00)00071-5. PMID 11068220
- [Background] Ilfeld BM. Continuous peripheral nerve blocks: a review of the published evidence. Anesth Analg. 2011 Oct;113(4):904-25. doi: 10.1213/ANE.0b013e3182285e01. Epub 2011 Aug 4. PMID 21821511
- [Background] Capdevila X, Ponrouch M, Choquet O. Continuous peripheral nerve blocks in clinical practice. Curr Opin Anaesthesiol. 2008 Oct;21(5):619-23. doi: 10.1097/ACO.0b013e32830c66c2. PMID 18784489
- Available data/document: Informed Consent Form — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisaAgrupador.jsf